CLINICAL TRIAL: NCT05118555
Title: Evaluation of New Magnetic Resonance Techniques
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5359
Record Dates: First submitted 2021-10-18; First posted 2021-11-12 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 1: Patients scheduled to undergo a routine clinical MR examination of the relevant anatomical regions and/or disease type will be identified from MRI department schedules.
  The new MR technique will be used to acquire additional data in patients undergoing a routine MR examination. The routine MR examination will be conducted according to the standard protocol.
- Type 2: Patients with the relevant disease type and no contraindications to MRI will be identified by delegated radiologists in clinics.
  An additional MR examination will be scheduled; this examination is in addition to any examinations that the patient may undergo as part of their clinical care. The MR examination will be conducted using the new MR technique; standard MR techniques may also be used for comparison.
- Type 3: Normal volunteers who are members of staff or students at RMH/ICR will be invited to participate using a mailing list. Exceptionally employees of other NHS Trusts and Academic Institutions will be allowed to participate if they are in collaboration with RMH/ICR.
  An MR examination will be conducted using the new MR technique; standard MR techniques may also be used for comparison.

SUMMARY:
The aim of this research protocol is to undertake evaluation of new and emerging MR techniques in patients and healthy volunteers following software or hardware upgrades, as well as for newly developed MR techniques; to establish their feasibility, image quality and/or measurement repeatability/ reproducibility.

DETAILED DESCRIPTION:
This study is a 'master protocol', analogous to an umbrella trial design, that seeks to evaluate multiple new MR techniques. As such, the study is designed to identify promising techniques that merit further investigation. Following successful evaluation as part of this study, new MR techniques will either be adopted into clinical practice or developed further in a larger research study.

Type 1) The new measurements are added to an existing patient examination, to allow evaluation of the benefits of the new approach in comparison with standard procedures, in the pathology of interest. This frequently is required during development of a new approach, when measurements indicate shortcomings that can be corrected by modification of the sequence, or in assessing a new software release from the manufacturer, which provides a range of new or improved facilities, that must be assessed in relation to our established approach. In this case patients undergoing established procedures or protocols will be measured with additional sequences provided that the additional examinations do not add more than 15 minutes to the total examination, that exposure is below or within the first level controlled MR safety mode, and is not indicated to be likely to cause any adverse effects. No additional intra-venous contrast agents will be administered (patients will receive intra-venous contrast agent if indicated as part of their routine examination). These measurements will be performed with verbal consent from the patient, which will be documented in the patient's Electronic Patient Record (EPR).

Type 2) The measurements for evaluation or development of a new technique (usually in a research setting) require a complete measurement or series of measurements to evaluate the technique in appropriate pathology, often during the course of treatment. These measurements will typically last for 30-60 minutes, the duration of standard MR examinations. In exceptional circumstances these measurements will last up to 90 minutes. Measurements will be conducted with the consent of the clinician responsible for the patient, which will be documented in the patient's Electronic Patient Record (EPR). Measurements will be performed with written informed consent from the patient. As this is a dedicated session for the purpose of evaluating the new technique, this will require informed consent with a clear indication of any potential adverse effects in the patient information sheet, even if such measurement is performed during a routine clinically indicated or research examination. No intra-venous contrast agents will be administered as a part of this protocol.

Type 3) The measurements for evaluation or development of a new technique require measurements in normal volunteers to establish the correct operation and value of the technique, and in some cases to assess measurement repeatability or reproducibility. These measurements will typically last for 30-60 minutes, the duration of standard MR examinations. In exceptional circumstances these measurements will last up to 90 minutes. Measurements will be performed with written informed consent from the volunteer. Any potential adverse effects will be clearly indicated in the volunteer information sheet. No intra-venous contrast agents will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Type 1: Patients undergoing a routine clinical MR examination using established MR techniques to which an additional new sequence is added for evaluation, who give verbal consent for additional data to be acquired for evaluation of a new MR technique.
* Type 2: Patients who voluntarily agree to participate in the study by giving written informed consent.
* Type 3: Normal volunteers who voluntarily agree to participate in the study by giving written informed consent.

Exclusion Criteria:

* Standard MR Exclusion criteria apply to all MR examinations, as documented in the MRI Local Rules.
* Patients or volunteers who are unwilling to undergo an additional MR examination, for example due to claustrophobia, will be excluded from the study.
* Normal volunteers who do not have an NHS number or who are not registered with a GP will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Royal Marsden Hospital patients and normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 2850 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a new MR technique | 10 years
  Assessment of feasibility is required at the earliest stages of development of a new MR technique. We will assess whether a new MR technique can be implemented on our MRI scanners with at least 60% success in achieving the desired measurement. 'Success' will be defined as: i. Acceptable quality of the MR image (or other MR data), assessed by a consultant radiologist or MR physicist, depending in the technique being investigated. ii. Acquisition time up to 15 minutes per sequence.
Qualitative assessment of a new MR technique (e.g. image quality) | 10 years
  mage quality will be assessed using a 5-point Likert scale (1 = unacceptable/non diagnostic images, 2 = diagnostic images with some artefacts affecting interpretation, 3 = moderate quality images, 4 = good, 5 = excellent image quality with no artefacts)
Objective comparison of a new MR technique with a current MR technique | 10 years
  (1 = unacceptable/non diagnostic images, 2 = diagnostic images with some artefacts affecting interpretation, 3 = moderate quality images, 4 = good, 5 = excellent image quality with no artefacts)
Assessment of repeatability or reproducibility of a quantitative metric using a new MR technique | 10 years
  Repeatability or reproducibility will be assessed using two measurements separated by a short time interval using the same MRI scanner (repeatability) or a different MRI scanner (reproducibility). Bland-Altman plots will be used to assess repeatability / reproducibility and 95% limits of agreement (LoA) will be estimated.
Assessment of a new MR technique in pre- and post-treatment measurements | 10 years
  Quantitative measurements from a new MR technique will be assessed in pre- and post treatment measurements, in order to assess the dynamic range of post-treatment changes relative to the repeatability of the measurement. These data will be used to assess whether further clinical studies are warranted for assessment of the new technique as a potential imaging biomarker. (The treatment is not part of this study, and will be standard-of-care. The timepoints will be defined relative to the standard-of-care pathway and will be fixed for all patients assessed per disease/MR technique.)

CONTACTS AND LOCATIONS:
Overall Officials: Dow-Mu Koh, MD,FRCP,FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Rata M, Castagnoli F, Shur J, Evans E, Hopkinson G, Benkert T, Weiland E, Koh DM, Winfield JM. Qualitative and quantitative assessment of accelerated liver diffusion-weighted imaging using deep-learning reconstruction in oncologic patients. BMC Med Imaging. 2025 Nov 26;25(1):491. doi: 10.1186/s12880-025-02030-3. PMID 41299300